CLINICAL TRIAL: NCT02708836
Title: Limiting Emergence Phenomena After General Anesthesia for Laparoscopic Surgery With Combined Laryngeal Mask Airway and Endotracheal Tube Airway Management Technique
Brief Title: Limiting Emergence Phenomena After General Anesthesia With Combined LMA and ETT Airway Management Technique
Acronym: LEPAGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Principal Investigator, Arne Budde, Associate Professor, Department of Anesthesiology and Perioperative Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 00004373
Record Dates: First submitted 2016-03-04; First posted 2016-03-15 (Estimated); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Limit Emergence Phenomena After General Anesthesia
MeSH Terms: interventions — Laryngoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ETT only (Active Comparator): Endotracheal tube intubation after induction of anesthesia. Ventilation with ETT until emergence.
  Interventions: Procedure: Induction of anesthesia; Device: Laryngoscopy and placement of ETT; Procedure: Ventilation via the ETT; Procedure: Removal of the ETT; Procedure: Emergence from anesthesia
- Combined ETT/LMA technique (Experimental): Placement of LMA after induction of anesthesia. Intubation of trachea with ETT via LMA with fiberoptic bronchoscope. Ventilation with ETT throughout case. Removal of ETT while deeply anesthetized. Ventilation with LMA until emergence.
  Interventions: Procedure: Induction of anesthesia; Device: Placement of LMA [Ambu (R) AuraGain (TM) disposable laryngeal mask]; Procedure: Ventilation via the ETT; Procedure: Removal of the ETT; Procedure: Intubation of the trachea through the LMA; Procedure: Ventilation via the LMA; Procedure: Emergence from anesthesia

INTERVENTIONS:
Procedure: Induction of anesthesia — At the discretion of the primary anesthesiologist. Typically involves the administration of an analgesic agent, hypnotic agent, and neuromuscular blocking agent
Device: Placement of LMA [Ambu (R) AuraGain (TM) disposable laryngeal mask] — By standard method. Sizing at the discretion of the primary anesthesiologist.
  Arms: Combined ETT/LMA technique
Device: Laryngoscopy and placement of ETT — Via direct or indirect laryngoscopy. Sizing at the discretion of the primary anesthesiologist. Mallinckrodt (TM) Intermediate Hi-Lo cuffed endotracheal tube (Covidien)
  Arms: ETT only
Procedure: Ventilation via the ETT — Ventilator mode, tidal volume/ ventilation pressure, respiratory rate, positive end expiratory pressure, inspired to expired ratio at the discretion of the primary anesthesiologist.
Procedure: Removal of the ETT — Either upon emergence of anesthesia after suctioning of the oropharynx and after a positive pressure breath or while deeply anesthetized after release of the pneumoperitoneum in the combined LMA/ETT group.
Procedure: Intubation of the trachea through the LMA — With ETT using fiberoptic bronchoscope guidance.
  Arms: Combined ETT/LMA technique
Procedure: Ventilation via the LMA — After removal of the ETT. Ventilator mode, tidal volume/ ventilation pressure, respiratory rate, positive end expiratory pressure, inspired to expired ratio at the discretion of the primary anesthesiologist.
  Arms: Combined ETT/LMA technique
Procedure: Emergence from anesthesia — At the discretion of primary team. Airway device (either ETT or LMA) will be removed when patient is adequately ventilating and able to respond to commands (such as "open your eyes" or "squeeze my hand").

SUMMARY:
Emergence from general anesthesia with a laryngeal mask airway compared with an endotracheal tube has been shown to favorable with respect to limiting emergence phenomena such as coughing, straining, restlessness, and sympathetic stimulation leading to hypertension and tachycardia.

Many anesthesiologists would prefer the use of an ETT to an LMA in cases in which higher ventilation pressures may be required, in those patients who are perceived to be high risk for reflux and pulmonary aspiration of gastric contents, as well as during cases that allow the anesthesiologist to have little accessibility the airway.

The aim of this study is to investigate an airway management technique that would allow for the benefits of the ETT in terms of a secure airway for the duration of the surgical procedure as well the potential for less emergence phenomena seen when emerging with an LMA.

DETAILED DESCRIPTION:
Emergence from general anesthesia is a critical period of anesthetic management (1. Popat, 2012). The noxious stimuli of an endotracheal tube as well as the excitement stage of anesthesia, commonly seen prior to return of consciousness while emerging from general anesthesia, both lead to emergence phenomena of coughing, straining, and restlessness in addition to physiologic derangements (2. Atkinson, 1987). Physiologically, emergence from anesthesia is associated with rising sympathetic tone (as evidenced by elevated catecholamine levels and the resultant hemodynamic changes of increasing heart rate and blood pressure), intracranial pressure, and intraocular pressure. Airway tone and reflexes are also problematic as they may be depressed by the lingering pharmacologic effects of anesthetics and analgesics leading to decreased airway obstruction or aspiration events. Airway reflexes may also be exaggerated while traversing the excitement stage; this can lead to undesirable consequences of coughing, breath-holding, bucking or in extreme cases laryngospasm. A smooth emergence is preferable for all patients but is required for those patients who would not tolerate the above physiologic changes (e.g. severe aortic stenosis or coronary artery disease, both of which would poorly tolerate tachycardia) or those would be at risk in terms of the procedure that was performed (cerebral aneurysm clipping, carotid endarterectomy, thyroidectomy: procedures in which stress fresh surgical wounds with hypertension and straining would be undesirable).

Several airway management (3. Koga 1998, 4. Perello-Cerda 2015) and pharmacologic strategies (5. Minogue 20014, 6. Nho 2009, 7. Guler 2005) have been employed to provide a smooth emergence from general anesthesia. One of the most efficacious strategies is the use of supraglottic airway devices rather than endotracheal tubes. Despite evidence supporting the safety and efficacy of ventilation of SGAs during laparoscopic procedures (8. Natalini 2003, 9. Belena 2012, 10. Carron 2012, 11. Bernardini 2009), many anesthesiologists would prefer the use of an ETT to an SGA in cases in which higher ventilation pressures may be required (obesity, steep Trendeleberg position, pneumoperitoneum). In addition to the cases requiring high ventilation pressures, ETTs are preferred to SGAs in those patients who are perceived to be high risk for reflux and pulmonary aspiration of gastric contents (non-fasted, intestinal obstruction, gastroparesis, parturients), as well as during cases that allow the anesthesiologist to have little accessibility the airway (neurosurgical, ENT, etc).

The Bailey maneuver (managing the airway with an ETT throughout the case and then exchanging for an LMA while deeply anesthetized (12. Nair 1995), has also been shown to provide less stimulating emergence. Unfortunately, the Bailey maneuver is relatively contraindicated in cases in which there is the perception that reintubation would be difficult, as the risks of exchanging a functioning airway device for one that has not been tested outweighs the potential benefits of a smooth emergence.

The airway management technique under investigation involves initially placing an LMA after induction of anesthesia. Once adequate ventilation has been accomplished using the LMA, the patient will be endotracheally intubated using a fiberoptic bronchoscope and the in situ LMA as a conduit (13. Timmermann 2011). General anesthesia will be maintained with sevoflurane and narcotics at the discretion of the primary anesthesiologist. The patient will be ventilated via the endotracheal tube during the duration of the surgical procedure and then the trachea will be extubated while the patient is at a deep plane of anesthesia after release of the pneumoperitoneum and return to supine positioning. This technique is a potential method for reducing the stress of emergence in patients who would benefit from the use of an endotracheal tube intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Patients undergoing elective laparoscopic surgery

Exclusion Criteria:

* Individuals who cannot provide consent
* Individuals who would require translation services to provide consent
* Prisoners
* Parturients
* Non-fasted patients (as per HMC Anesthesiology Department NPO policy)
* Patients felt to be high risk for gastric reflux and pulmonary aspiration (those with gastroparesis, symptomatic GERD, etc.: at the discretion of primary anesthesia team) Those patients with anticipated difficult airway requiring maintenance of spontaneous ventilation (awake intubation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in rate pressure product during emergence | Intraoperative
  Difference in heart rate multiplied by systolic blood pressure measured during the ~5 minutes prior to emergence and the ~5 minutes after removal of the airway device. Heart rate is continuously monitored and recorded at one minute intervals. Blood pressure is intermittently monitored at 3 minute intervals. The two SBPs measured prior to removal of the airway device will be multiplied by the HR at those times and the RPPs will be averaged. This will be compared with average of the product of the two SBPs and their corresponding HRs measured after removal of the airway device.

SECONDARY OUTCOMES:
Time to successful ventilation via ETT | Intraoperative
  From administration of induction medication until ETT placement confirmed via capnography.
Change in rate pressure product during induction of anesthesia and intubation | Intraoperative
  Difference in heart rate multiplied by systolic blood pressure measured during the ~5 minutes prior to induction of anesthesia and the ~5 minutes after placement of the airway device. Heart rate is continuously monitored and recorded at one minute intervals. Blood pressure is intermittently monitored at 3 minute intervals. The two SBPs measured prior to placement of the airway device will be multiplied by the HR at those times and the RPPs will be averaged. This will be compared with average of the product of the two SBPs and their corresponding HRs measured after placement of the airway device.
Success rate of ventilation with LMA after extubation of trachea | Intraoperative
  After deflation of the pneumoperitoneum, the ETT will be removed and ventilation will be continued through the LMA.
  Success will be graded as follows:
  1. Adequate ventilation via LMA without need for adjustment.
  2. Adequate ventilation via LMA after adjustment of LMA.
  3. Inadequate ventilation via LMA. Unable to successfully re-seat LMA and need to re-intubate.
Presence/ severity of cough during prior to removal of airway device | Intraoperative
  During 5 minutes prior to removal of airway device.
  Cough will be graded as follows:
  None Mild = 1 episode of unsustained coughing (< 5 s) Moderate = More than 1 episode of unsustained (<5 s) coughing Severe = Sustained bout(s) of coughing (>5 s) http://www.ncbi.nlm.nih.gov/pubmed/15385385 - (5. Minogue 2004)
Presence/ severity of cough during after removal of airway device | Intraoperative
  During 5 minutes after removal of airway device.
  Cough will be graded as follows:
  None Mild = 1 episode of unsustained coughing (< 5 s) Moderate = More than 1 episode of unsustained (<5 s) coughing Severe = Sustained bout(s) of coughing (>5 s) http://www.ncbi.nlm.nih.gov/pubmed/15385385 - (5. Minogue 2004)
Total opioids (morphine equivalents) administered intraoperatively | Intraoperative
  From pre-induction until patient hand-off to post-anesthesia care unit team. Total intraoperative narcotics will be converted to morphine equivalents.
LMA cuff pressures when inflated to seal | Intraoperative
  After placement of LMA and LMA cuff inflated to seal. Pressure in the cuff will be measured and then deflated to pressures of 50-60 cmH20.
LMA cuff pressures prior to removal of ETT. | Intraoperative
  After deflation of the pneumoperitoneum. Pressure in the cuff will be measured and then deflated to pressures of 50-60 cmH20.
Presence of oropharyngeal sensory or motor nerve palsy. | Up to 1 week
  Postoperative day 3-5. A phone call will be made to determine the number of participants with the presence of any oropharyngeal numbness / paresthesias, hoarseness (recurrent laryngeal n. - Lehnert, 2008), dysphagia/ dysarthria (hypoglossal n. - Takahoko, 2014 & Shah, 2015), decreased sensation and sense of taste (lingual n. - El Toukhy, 2012) that could be indicative of a neuropraxia versus nerve palsy.
Presence of sore throat. | Up to 1 week
  Postoperative day 3-5. A phone call will be made to determine the number of participants with sore throat (subjectively rated as none, mild, or severe).

CONTACTS AND LOCATIONS:
Overall Officials: Arne Budde, MD, Principal Investigator — Penn State M.S. Hershey Medical Center
Locations (1):
- Penn State Health - Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be stored in REDCap, a HIPPA compliant secured and encrypted electronic database.

REFERENCES:
- [Result] Difficult Airway Society Extubation Guidelines Group; Popat M, Mitchell V, Dravid R, Patel A, Swampillai C, Higgs A. Difficult Airway Society Guidelines for the management of tracheal extubation. Anaesthesia. 2012 Mar;67(3):318-40. doi: 10.1111/j.1365-2044.2012.07075.x. PMID 22321104
- [Result] Atkinson RS, Rushman GB, Alfred Lee J: A Synopsis of Anaesthesia, 10th edition. Butterworth-Heinemann Ltd, 1987, pp 165-9
- [Result] Koga K, Asai T, Vaughan RS, Latto IP. Respiratory complications associated with tracheal extubation. Timing of tracheal extubation and use of the laryngeal mask during emergence from anaesthesia. Anaesthesia. 1998 Jun;53(6):540-4. doi: 10.1046/j.1365-2044.1998.00397.x. PMID 9709138
- [Result] Perello-Cerda L, Fabregas N, Lopez AM, Rios J, Tercero J, Carrero E, Hurtado P, Hervias A, Gracia I, Caral L, de Riva N, Valero R. ProSeal Laryngeal Mask Airway Attenuates Systemic and Cerebral Hemodynamic Response During Awakening of Neurosurgical Patients: A Randomized Clinical Trial. J Neurosurg Anesthesiol. 2015 Jul;27(3):194-202. doi: 10.1097/ANA.0000000000000108. PMID 25121397
- [Result] Minogue SC, Ralph J, Lampa MJ. Laryngotracheal topicalization with lidocaine before intubation decreases the incidence of coughing on emergence from general anesthesia. Anesth Analg. 2004 Oct;99(4):1253-1257. doi: 10.1213/01.ANE.0000132779.27085.52. PMID 15385385
- [Result] Nho JS, Lee SY, Kang JM, Kim MC, Choi YK, Shin OY, Kim DS, Kwon MI. Effects of maintaining a remifentanil infusion on the recovery profiles during emergence from anaesthesia and tracheal extubation. Br J Anaesth. 2009 Dec;103(6):817-21. doi: 10.1093/bja/aep307. Epub 2009 Oct 28. PMID 19864308
- [Result] Guler G, Akin A, Tosun Z, Eskitascoglu E, Mizrak A, Boyaci A. Single-dose dexmedetomidine attenuates airway and circulatory reflexes during extubation. Acta Anaesthesiol Scand. 2005 Sep;49(8):1088-91. doi: 10.1111/j.1399-6576.2005.00780.x. PMID 16095449
- [Result] Natalini G, Lanza G, Rosano A, Dell'Agnolo P, Bernardini A. Standard Laryngeal Mask Airway and LMA-ProSeal during laparoscopic surgery. J Clin Anesth. 2003 Sep;15(6):428-32. doi: 10.1016/s0952-8180(03)00085-0. PMID 14652119
- [Result] Beleña JM, Núñez M, Gracia JL, Pérez JL, Yuste J. The Laryngeal Mask Airway Supreme™: safety and efficacy during gynaecological laparoscopic surgery. Southern African Journal of Anaesthesia and Analgesia 18: 143-7, 2012.
- [Result] Carron M, Veronese S, Gomiero W, Foletto M, Nitti D, Ori C, Freo U. Hemodynamic and hormonal stress responses to endotracheal tube and ProSeal Laryngeal Mask Airway for laparoscopic gastric banding. Anesthesiology. 2012 Aug;117(2):309-20. doi: 10.1097/ALN.0b013ef31825b6a80. PMID 22614132
- [Result] Bernardini A, Natalini G. Risk of pulmonary aspiration with laryngeal mask airway and tracheal tube: analysis on 65 712 procedures with positive pressure ventilation. Anaesthesia. 2009 Dec;64(12):1289-94. doi: 10.1111/j.1365-2044.2009.06140.x. Epub 2009 Oct 23. PMID 19860753
- [Result] Nair I, Bailey PM. Use of the laryngeal mask for airway maintenance following tracheal extubation. Anaesthesia. 1995 Feb;50(2):174-5. doi: 10.1111/j.1365-2044.1995.tb15104.x. No abstract available. PMID 7710032
- [Result] Timmermann A. Supraglottic airways in difficult airway management: successes, failures, use and misuse. Anaesthesia. 2011 Dec;66 Suppl 2:45-56. doi: 10.1111/j.1365-2044.2011.06934.x. PMID 22074079
- [Result] Takahoko K, Iwasaki H, Sasakawa T, Suzuki A, Matsumoto H, Iwasaki H. Unilateral hypoglossal nerve palsy after use of the laryngeal mask airway supreme. Case Rep Anesthesiol. 2014;2014:369563. doi: 10.1155/2014/369563. Epub 2014 Aug 31. PMID 25254120
- [Result] Lehnert B, Prescher A, Neuschaefer-Rube C. Is laryngeal mask airway-related vocal chord palsy always laryngeal mask airway-related? Br J Anaesth. 2008 Dec;101(6):882. doi: 10.1093/bja/aen304. No abstract available. PMID 19004921
- [Result] El Toukhy M, Tweedie O. Bilateral lingual nerve injury associated with classic laryngeal mask airway: a case report. Eur J Anaesthesiol. 2012 Aug;29(8):400-1. doi: 10.1097/EJA.0b013e3283514e81. No abstract available. PMID 22472625
- [Result] Shah AC, Barnes C, Spiekerman CF, Bollag LA. Hypoglossal nerve palsy after airway management for general anesthesia: an analysis of 69 patients. Anesth Analg. 2015 Jan;120(1):105-120. doi: 10.1213/ANE.0000000000000495. PMID 25625257